CLINICAL TRIAL: NCT02858414
Title: Exploratory Study of Cellular Reservoirs in Blood From HIV Infected Patients: EURECA (ERANET to Unravel New Roads to Eradication and a Cure for AIDS) Study
Brief Title: Exploratory Study of Cellular Reservoirs in Blood From HIV Infected Patients
Acronym: EURECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P/2014/223
Record Dates: First submitted 2016-07-29; First posted 2016-08-08 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- blood sample (Experimental)
  Interventions: Other: additional blood sample

INTERVENTIONS:
Other: additional blood sample

SUMMARY:
This study evaluates the impact of highly active antiretroviral therapy on the size of the latent viral reservoirs in resting CD4+ T cells and monocytes in HIV positive patients. The activation state of the cells will be assessed, by measuring the activation of Akt, to determine its influence on the size of the viral reservoirs.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients under Highly Active Anti-Retroviral Therapy (HAART) or Naïve from treatment

Exclusion Criteria:

* Age limits
* Pregnancy
* Legal restrictions to consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Measure of the integrated viral reservoir size | day 1
  Measure by Alu-PCR. Results are given in number of integrated proviral DNA copies per 1 million cells.
Measure of the proviral reservoir size | day 1
  Measure by Total Proviral HIV DNA detection kit. Results are given in number of total proviral DNA copies per 1 million cells.

SECONDARY OUTCOMES:
Measure of Akt activation | day 1
  Measure of Akt activation in live cells by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Georges HERBEIN, MD-PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- Centre Hospitalier Régional Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No